CLINICAL TRIAL: NCT01779882
Title: Cyclophosphamide-Busulfan Versus Busulfan-Cyclophosphamide as Conditioning Regimen Before Allogeneic Hematopoietic Stem Cell Transplantation for Leukemia: a Prospective Randomized Study to Assess Liver Toxicity
Brief Title: Cyclophosphamide and Busulfan as Conditioning Regimen Before Allogeneic HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Zürich (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BuCyBu study
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Myeloid Leukemia; Precursor Myeloid Neoplasms; Lymphoid Neoplasms
MeSH Terms: conditions — Leukemia, Myeloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BU-CY (Active Comparator): Group A (standard group): conditioning regimen with Busulfan (BU) followed by Cyclophosphamide (CY)
  Interventions: Drug: Busulfan-Cyclophosphamide as Conditioning Regimen before Allogeneic Hematopoietic Stem Cell Transplantation
- CY-BU (Experimental): Group B (experimental group): conditioning regimen with Cyclophosphamide (CY) followed by Busulfan (BU)
  Interventions: Drug: Cyclophosphamide-Busulfan as Conditioning Regimen before Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: Busulfan-Cyclophosphamide as Conditioning Regimen before Allogeneic Hematopoietic Stem Cell Transplantation — Test the hypothesis, that the order of application of Busulfan (BU) and Cyclophosphamide (CY) has an impact on toxicity after allogeneic Hematopoietic stem cell transplantation (HSCT) and that CY-BU reduces liver toxicity compared to BU-CY.
  Arms: BU-CY
Drug: Cyclophosphamide-Busulfan as Conditioning Regimen before Allogeneic Hematopoietic Stem Cell Transplantation — Test the hypothesis, that the order of application of Busulfan (BU) and Cyclophosphamide (CY) has an impact on toxicity after allogeneic Hematopoietic stem cell transplantation (HSCT) and that CY-BU reduces liver toxicity compared to BU-CY.
  Arms: CY-BU

SUMMARY:
The aim of this study is to test the hypothesis, that the order of application of Busulfan (BU) and Cyclophosphamide (CY) has an impact on toxicity after allogeneic Hematopoietic stem cell transplantation (HSCT) and that CY-BU reduces liver toxicity compared to BU-CY.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo an allogeneic HSCT with myeloablative conditioning
* Age 18 - 65 years
* Myeloid leukemia respectively related precursor neoplasms (acute myeloid leukemia, chronic myeloid leukemia, myelodysplastic syndrome), or lymphoid neoplasms (acute lymphoblastic leukemia/lymphoma, mature B-/T-/natural killer (NK)-cell neoplasms).
* Human Leukocyte Antigen (HLA)-identical sibling donor or matched unrelated (min. 10/10 Ag matched)
* Patients with a history of hepatitis might be included, if no contraindication for HSCT exists.
* Patient must give written informed consent

Exclusion Criteria:

* Indication other than myeloid leukemia respectively related precursor neoplasms, or lymphoid neoplasms.
* Severe liver damage for > 2 weeks (bilirubin > 3xupper limit normal (ULN) or ASAT/ALAT > 5xULN)
* HIV infection
* Donor other than HLA-identical sibling or min. 10/10 matched unrelated donor
* Pregnant or lactating women
* Lack of written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2018-01-06 (Actual); Study Completion 2018-01-06 (Actual)

PRIMARY OUTCOMES:
Liver toxicity | Day 30
  Liver toxicity, assessed as absolute serum values of ASAT, ALAT, GGT, Alkaline Phosphatase, bilirubin at day 30.

SECONDARY OUTCOMES:
VOD | Day 30
  Incidence and severity of "veno occlusive disease (VOD)" at day 30
Acute graft-versus-host disease (GvHD) | Day 30 and Day 100
  Incidence and severity of acute GVHD, by organ (skin, liver, gut) at day 30 and day 100
Toxicity | Day 30 and Day 100
  Organ toxicity at day 30 and day 100
Efficacy | Day 30 and Day 100
  Survival, relapse and non-relapse mortality at day 30 and day 100
Cumulative liver values | Day 0, 10, 20 and 30
  Cumulative serum values of aspartate transaminase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyltransferase (GGT), Alkaline Phosphatase, bilirubin for days 0, 10, 20 and 30
Maximum liver values | Day 0, 10, 20 and 30
  Maximum serum values of ASAT, ALAT, GGT, alkaline phosphatase (AP), bilirubin at any time between day 0 and day 30

OTHER OUTCOMES:
Cytokines measurement | Day -8, 0, 10, 20 and 30
  To test the correlation between order of application of the conditioning regimen and the levels of proinflammatory cytokines as well as the correlation between levels of cytokines and development of acute GVHD, plasma samples will be collected at different time points.
Pharmacogenomics | Day -8, -3 and 0
  The current hypothesis is that some functional polymorphisms of genes, which control important enzymes in BU and CY metabolism, contribute to the observed interindividual variability in toxicity after allogeneic HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Cantoni, MD, Study Chair — Kantonsspital Aarau, Switzerland; Sabine Gerull, MD, Principal Investigator — University Hospital, Basel, Switzerland; Gayathri Nair, MD, Principal Investigator — University Hospital, Zürich; Yves Chalandon, MD, Principal Investigator — University Hospital Geneva, Switzerland; Jakob Passweg, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - University Hospital, Basel, Basel
  - University Hospital Geneva, Geneva
  - University Hospital Zurich, Zurich

REFERENCES:
- [Background] Cantoni N, Gerull S, Heim D, Halter J, Bucher C, Buser A, Tsakiris DA, Passweg J, Tichelli A, Stern M, Gratwohl A. Order of application and liver toxicity in patients given BU and CY containing conditioning regimens for allogeneic hematopoietic SCT. Bone Marrow Transplant. 2011 Mar;46(3):344-9. doi: 10.1038/bmt.2010.137. Epub 2010 Jun 14. PMID 20548339
- [Derived] Seydoux C, Uppugunduri CRS, Medinger M, Nava T, Halter J, Heim D, Chalandon Y, Schanz U, Nair G, Cantoni N, Passweg JR, Ansari M. Effect of pharmacokinetics and pharmacogenomics in adults with allogeneic hematopoietic cell transplantation conditioned with Busulfan. Bone Marrow Transplant. 2023 Jul;58(7):811-816. doi: 10.1038/s41409-023-01963-z. Epub 2023 Apr 21. PMID 37085674